CLINICAL TRIAL: NCT02332499
Title: Randomized,Double-blind,Placebo-controlled,Multicenter Study to Compare the Efficacy and Safety of Anlotinib Plus BSC Versus Placebo Plus BSC in Patients With Metastatic Colorectal Cancer Refractory to Standard Chemotherapies(ALTER0703)
Brief Title: Study of Anlotinib in Patients With Metastatic Colorectal Cancer（mCRC）(ALTER0703)
Acronym: ALTER0703
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-07-IIB
Record Dates: First submitted 2014-12-31; First posted 2015-01-06 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Anlotinib; Metastatic Colorectal Cancer （mCRC）; ALTER0703
MeSH Terms: conditions — Colorectal Neoplasms | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anlotinib (Active Comparator): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib
- Placebo (Placebo Comparator): Placebo QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anlotinib — Anlotinib p.o. qd
  Other Names: AL3818
  Arms: Anlotinib
Drug: Placebo — Placebo p.o. qd
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effects and safety of Anlotinib with placebo in patients with metastatic colorectal cancer refractory to standard chemotherapies.

DETAILED DESCRIPTION:
Anlotibib (AL3818) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA:2011L00661） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd.To compare the effects and safety of Anlotinib with placebo in patients with metastatic colorectal cancer refractory to standard chemotherapies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent；
2. Histological or cytological documentation of adenocarcinoma of the colon or rectum；
3. Subjects with metastatic colorectal cancer (Stage IV),With measurable disease (using RECIST1.1)；
4. Progression during or within 3 months following the last administration of approved standard therapies which must include Fluorouracil or its derivatives, Oxaliplatin, Irinotecan；
5. ECOG PS:0-1,Life expectancy of more than 3 months；
6. main organs function is normal；
7. main organs function is normal；

Exclusion Criteria:

1. Prior treatment with Anlotinib；
2. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study drug；
3. Known brain metastases；
4. patients with severe and failed to controlled diseases；
5. patients occurred venous thromboembolic events within 6 months；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08-18 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)

SECONDARY OUTCOMES:
Progress free survival (PFS) | each 42 days up to PD or death(up to 24 months)
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Until 30 day safety follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Yihebali Chi, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jianqiang Cai, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jinwan Wang, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (29):
- China (29):
  - The 1st Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Second Affiliated Hospital, Anhui Medical University, Hefei, Anhui
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The 307th Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Gansu Province Tumor Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Sun Yat-sen university, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen university, Guangzhou, Guangdong
  - Guangxi medical university affiliated tumor hospital, Nanning, Guangxi
  - Harbin medical university affiliated tumor hospital, Haerbin, Heilongjiang
  - The Second xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Cancer Hospital, Nantong, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Province Tumor Hospital, Shenyang, Liaoning
  - Qilu Hospital，Shandong University, Jinan, Shandong
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Xian, Shanxi
  - Tangdu Hospital of The fourth Military Medical University, Xian, Shanxi
  - The First Affiliated Hospital of Xian Jiaotong University, Xian, Shanxi
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- See also: Cancer — http://www.nlm.nih.gov/medlineplus/cancer.html
- See also: Colorectal Cancer — http://www.nlm.nih.gov/medlineplus/colorectalcancer.html
- See also: U.S. FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks